CLINICAL TRIAL: NCT03003403
Title: Balance: A Pragmatic Trial of a Digital Health Intervention to Prevent Weight Gain in Primary Care
Acronym: D0479
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0738
Record Dates: First submitted 2016-12-16; First posted 2016-12-28 (Estimated); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Overweight; Overnutrition; Nutrition Disorders; Signs and Symptoms
Keywords: mHealth; Digital Health; Primary Care; Pragmatic Clinical Trial; Behavior Change; Weight Management
MeSH Terms: conditions — Obesity; Overweight; Overnutrition; Nutrition Disorders; Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Program (Experimental): Balance Intervention Program: Participants randomly assigned to the 12-month digital health behavioral intervention will receive: tailored behavior change goals with interactive self-monitoring and feedback; network-connected scales to track their weight; skills training materials; and stepped coaching (via phone and/or text) from Registered Dieticians serving as health coaches within a local network of community health centers.
  Interventions: Behavioral: Intervention Program
- Usual Care Program (No Intervention): Balance Usual Care Program: Participants randomly assigned to the Usual Care program will receive the standard primary care offered by their providers; health information/skills training materials to maintain a healthy weight; and automated (non-tailored) text messages with health information.

INTERVENTIONS:
Behavioral: Intervention Program — Balance is testing a pragmatic approach to promote weight maintenance among overweight patients and patients with obesity within local community health centers who experience barriers to losing weight. The intervention utilizes the interactive obesity treatment approach, which creates an energy deficit by having participants achieve simple, straightforward, and concrete behavior change goals (e.g., no fast food, no sugary drinks, walk 10,000 steps per day). The Balance intervention involves tailored behavior change goals; self-monitoring using connected scales and mobile technologies; responsive coaching, and tailored feedback and skills training.
  Arms: Intervention Program

SUMMARY:
Up to 50% of obese patients are not interested in, or ready for, weight loss. Clinical practice guidelines clearly recommend that these patients avoid gaining weight. However, despite this clinical guideline, weight gain prevention interventions are not available in primary care practice. Balance is a pragmatic, randomized controlled effectiveness trial for weight gain prevention for patients within rural community health centers, using a digital health platform.

DETAILED DESCRIPTION:
Clinical practice guidelines emphasize recommend weight gain prevention, but evidence-based treatments are not available in primary care. Balance, a pragmatic effectiveness trial, will test a scalable treatment approach for medically-vulnerable adults, those who suffer disproportionately from obesity and its adverse health effects. Balance builds on the design and findings of the Shape study (NCT00938535) to test a pragmatic intervention within rural community health centers. Balance will randomize overweight adults and adults with obesity who are patients a local community health center network (Piedmont Health Services) to either: 1) a 12-month weight gain prevention intervention or 2) usual care. Intervention group components include tailored behavior change goals; mHealth self-monitoring and feedback; skills training videos; and stepped responsive coaching from clinic Registered Dietitians. The usual care group will receive standard primary care offered by their providers and automated text messages and health information about maintaining a healthy weight. All intervention components and materials will be provided in Spanish or English.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Piedmont Health Services' community health centers in central North Carolina only
* BMI between 25 and 40 kg/m2 and weighs less than 380 lbs
* Speaks English or Spanish
* Had a non-urgent outpatient visit at a participating community health center clinic at Piedmont Health Services within the last 2 weeks
* Has a cell phone
* Willing to receive 3-12 study-related text messages per week

Exclusion Criteria:

* Current Piedmont Health Services employee
* Has past bariatric surgery or planned bariatric surgery (within next 2 years)
* Diagnosed with cancer in the last 6 months and is in active treatment
* Has a history of cardiovascular event (stroke/MI) in the last 12 months
* Was hospitalized for a mental health issue in the last 12 months
* Diagnosis of end stage renal disease
* Currently participating in a weight loss program/research study
* Plans to move out of area and not receive care within community health center network (within the next 2 years)
* Currently or recently pregnant (within the last 6 months) - Females only
* Currently or recently lactating (with the last 2 months)- Females only
* Plans to get pregnant in the next 12 months - Females only

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary G Bennett, PhD, Principal Investigator — Duke University; Dori M Steinberg, PhD, RD, Principal Investigator — Duke University
Locations (1):
- Duke University - with Piedmont Health Services, Inc., Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller HN, Gallis JA, Askew S, Lee A, Berger MB, Kay MC, Egger JR, Bennett GG. Assessing Electronic Health Record-Derived Outcomes in a Pragmatic Weight Gain Prevention Trial: Effects, Variability, and Implications for Future Trials. J Cardiovasc Nurs. 2026 Mar-Apr 01;41(2):E57-E62. doi: 10.1097/JCN.0000000000001281. Epub 2026 Jan 28. PMID 41603635
- [Derived] Miller HN, Gallis JA, Berger MB, Askew S, Egger JR, Kay MC, Finkelstein EA, de Leon M, DeVries A, Brewer A, Holder MG, Bennett GG. Weight Gain Prevention Outcomes From a Pragmatic Digital Health Intervention With Community Health Center Patients: Randomized Controlled Trial. J Med Internet Res. 2024 Mar 28;26:e50330. doi: 10.2196/50330. Erratum In: J Med Internet Res. 2024 May 13;26:e60137. doi: 10.2196/60137. PMID 38416574
- [Derived] Berger MB, Chisholm M, Miller HN, Askew S, Kay MC, Bennett GG. "We bleed for our community:" A qualitative exploration of the implementation of a pragmatic weight gain prevention trial from the perspectives of community health center professionals. BMC Public Health. 2023 Apr 14;23(1):695. doi: 10.1186/s12889-023-15574-2. PMID 37060053
- [Derived] Berger MB, Steinberg DM, Askew S, Gallis JA, Treadway CC, Egger JR, Kay MC, Batch BC, Finkelstein EA, DeVries A, Brewer A, Bennett GG. The Balance protocol: a pragmatic weight gain prevention randomized controlled trial for medically vulnerable patients within primary care. BMC Public Health. 2019 May 17;19(1):596. doi: 10.1186/s12889-019-6926-7. PMID 31101037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from partnering community health centers (CHCs) that worked with the Duke research team. Per privacy regulations, prior to being contacted by a team member, CHC patients were asked to review/sign a HIPAA authorization form to give permission to be contacted for recruitment. Once the form was received, study team members conducted an eligibility review in the CHC EHR. If eligible and interested, additional screening, verbal consent and randomization occurred via phone.
Pre-assignment Details: 443 participants were randomized after being eligible upon EHR chart review; phone screen and verbal consent and randomization.
Groups:
- Intervention Program: Balance Intervention Program: Participants randomly assigned to the 12-month digital health behavioral intervention will receive: tailored behavior change goals with interactive self-monitoring and feedback; network-connected scales to track their weight; skills training materials; and stepped coaching (via phone and/or text) from Registered Dietitians serving as health coaches within a local network of community health centers.
  Intervention Program: Balance is testing a pragmatic approach to promote weight maintenance among overweight patients and patients with obesity within local community health centers who experience barriers to losing weight. The intervention utilizes the interactive obesity treatment approach, which creates an energy deficit by having participants achieve simple, straightforward, and concrete behavior change goals (e.g., no fast food, no sugary drinks, walk 10,000 steps per day). The Balance intervention involves tailored behavior change goals; self-monitoring using connected scales and mobile technologies; responsive coaching, and tailored feedback and skills training.
Period: Overall Study
Arm/Group | Intervention Program | Usual Care Program
Started | 223 | 220
Completed | 212 | 212
Not Completed | 11 | 8
Not completed — Ineligible | 8 | 7
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Population: Final randomized sample was 443 participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Program | Usual Care Program | Total
Number analyzed (Participants) | 223 | 220 | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (13.6) | 46.8 (13.0) | 47.6 (13.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 43 | 46 | 89
  Female | 179 | 173 | 352
  Male to Female Transgender | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic (all races) | 102 | 98 | 200
  Non-Hispanic White | 61 | 54 | 115
  Non-Hispanic Black | 53 | 53 | 106
  Non-Hispanic other/unreported | 7 | 15 | 22
BMI [Mean (Standard Deviation); unit: kg/m2] | 32.4 (4.0) | 32.9 (3.9) | 32.6 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight at 24-months
Description: The proportion of intervention arm participants who achieve weight again prevention (staying within 3% of baseline weight in kg) at 24 months post-randomization. This will be calculated as follows: ((baseline weight in kg - final weight at 24 months in kg)/baseline weight in kg))x 100
Time Frame: Baseline, 24 months post-randomization (up to 27 months to obtain 24 month data)
Population: Entire sample analyzed for primary endpoint at 24-months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Program | Usual Care Program
Number analyzed (Participants) | 223 | 220
Participants
  Gained more than 3% | 28 | 29
  Gained less than or equal to 3% of predicted baseline weight | 88 | 90
  Not measured in time window | 107 | 101
Statistical Analysis 1: Comparison: Intervention Program vs Usual Care Program; Test type: Superiority; p = 0.97, bootstrap resampling; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.82 to 1.20]

2. Secondary Outcome: Change in Weight
Description: Average change in participant weight at 24 months post randomization, as measured in kg
Time Frame: Baseline, 24 months post-randomization (up to 27 months to obtain 24 month data)
Population: Average weight change (kg) at 24 months.
Measure: Mean (95% Confidence Interval); unit: change in weight by kg
Arm/Group | Intervention Program | Usual Care Program
Number analyzed (Participants) | 223 | 220
change in weight by kg | 0.4 [-0.4 to 1.2] | 0.5 [-0.3 to 1.5]
Statistical Analysis 1: Comparison: Intervention Program vs Usual Care Program; Test type: Superiority; p = 0.83, Mixed Models Analysis; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-1.24 to 1.00]

3. Secondary Outcome: Change in Blood Pressure
Description: Average change in participant systolic and diastolic blood pressure at 24 months post-randomization, as measured in millimeters of mercury (mm Hg), by arm
Time Frame: baseline, 24 months post-randomization (up to 27 months to obtain 24 month data)
Population: Predicted mean change (in mmHg) in systolic blood pressure and diastolic blood pressure, from baseline to 24 months, by study arm
Measure: Mean (95% Confidence Interval); unit: millimeters of mercury (mmHg)
Arm/Group | Intervention Program | Usual Care Program
Number analyzed (Participants) | 223 | 220
millimeters of mercury (mmHg)
  Average change in systolic blood pressure | -1.3 [-3.1 to 0.6] | -0.1 [-2 to 1.9]
  Average change in diastolic blood pressure | -2.8 [-4 to -1.5] | -2 [-3.3 to -0.7]
Statistical Analysis 1: Comparison: Intervention Program vs Usual Care Program; Test type: Superiority — Difference in systolic blood pressure change post-baseline comparing intervention to usual care arm at 24 months; p = 0.34, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-3.6 to 1.3]
Statistical Analysis 2: Comparison: Intervention Program vs Usual Care Program; Test type: Superiority — Difference in diastolic blood pressure change post-baseline comparing intervention to usual care arm at 24 months; p = 0.323, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.4 to 0.8]

4. Secondary Outcome: Change in Framingham Risk Score
Description: Average change in participant Framingham risk score at 24 months post-randomization, as measured by calculated 10-year Framingham risk score from the Framingham Heart Study. The Framingham Risk Score provides an estimate of the 10-year risk of developing cardiovascular disease. A decrease (negative) in score indicated a decreased 10-year risk of developing cardiovascular disease; an increase (positive) in score meant an increased 10-year risk of developing cardiovascular disease. Framingham score ranges vary by gender. For men, the minimum score is: -10 and maximum score is 21. For women: the min score is -8 and max score is 27.
Time Frame: baseline, 24 months post-randomization (up to 27 months to obtain 24 month data)
Population: Calculated mean change in 10-year cardiovascular risk between baseline and 24-months post-randomization by treatment arm.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Program | Usual Care Program
Number analyzed (Participants) | 223 | 220
units on a scale | -0.01 [-0.6 to 0.6] | -0.01 [-0.7 to 0.6]
Statistical Analysis 1: Comparison: Intervention Program vs Usual Care Program; Test type: Superiority; p = 0.991, Mixed Models Analysis; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-0.8 to 0.8]

ADVERSE EVENTS:
Time Frame: Randomization through 12 months (active intervention phase)
Description: We used the clinicaltrials.gov definitions for adverse events. Adverse events were collected directly from participants (email, phone, and/or text) and via medical chart reviews at 6- and 12-months.
Arm/Group | Intervention Program | Usual Care Program
All-Cause Mortality (participants affected / at risk) | 0/223 | 0/220
Serious Adverse Events (participants affected / at risk) | 22/223 | 13/220
Other Adverse Events (participants affected / at risk) | 42/223 | 34/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Program (N=223) | Usual Care Program (N=220)
Severe abdominal pain, discomfort, symptoms (Gastrointestinal disorders) | 3 (3) | 2 (2)
Motor vehicle accident; fall (Injury, poisoning and procedural complications) | 3 (3) | 0
Bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Cysts/Polyps requiring cancer treatment/other intervention (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Parkinson's related complications (Nervous system disorders) | 1 (1) | 2 (2)
Breathing complications (asthma, COVID19, infections) (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Surgical procedures for heart/GI (Surgical and medical procedures) | 1 (1) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1) | 0
Diabetes related complications (Endocrine disorders) | 1 (1) | 0
Kidney and urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Hypertension-related complications (Cardiac disorders) | 5 (5) | 4 (4)
Skin infections (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
General infectious diseases (Infections and infestations) | 2 (2) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Program (N=223) | Usual Care Program (N=220)
Hypertension-related issues (Cardiac disorders) | 5 (5) | 5 (5)
Minor falls (Injury, poisoning and procedural complications) | 11 (11) | 4 (4)
Eye infections (Eye disorders) | 3 (3) | 1 (1)
Minor UTIs (Renal and urinary disorders) | 4 (5) | 1 (1)
Minor stomach pain (Gastrointestinal disorders) | 4 (7) | 7 (7)
Sprains/strains (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (10)
Minor nerve pain/issues (Nervous system disorders) | 1 (2) | 1 (3)
Neoplasms/cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 (4)
Psychiatric condition (due to lack of medication) (Psychiatric disorders) | 0 | 1 (1)
Shortness of breath, minor respiratory infections (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 5 (6)
Uterine fibroid (Reproductive system and breast disorders) | 0 | 1 (1)
Diabetes-related complications (Endocrine disorders) | 1 (1) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0
Minor outpatient surgical procedures (Surgical and medical procedures) | 3 (3) | 0
Ear infection (Ear and labyrinth disorders) | 1 (1) | 0
Misc non-systemic infections (Infections and infestations) | 2 (2) | 0
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT03003403/Prot_SAP_ICF_000.pdf